CLINICAL TRIAL: NCT00450762
Title: Gemcitabine Plus Carboplatin in Patients With Pretreated Metastatic Breast Cancer
Brief Title: Gemcitabine + Carboplatin in Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Gem/Carbo MUC01
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Last update posted 2007-03-22 (Estimated); Status verified 2007-03

CONDITIONS: Breast Cancer
Keywords: pretreated; metastatic
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Gemcitabine; Carboplatin

INTERVENTIONS:
Drug: gemcitabine
Drug: carboplatin

SUMMARY:
The rational for this trial is given by the knowledge that gemcitabine acts as a potent inhibitor of DNA repair and therefore may prevent adequate repair of platin-induced DNA damage. Gemcitabine is an excellent choice for combination therapy by its unique mechanism of action and favourable toxicity profile. The combination of gemcitabine and cisplatin was shown to be effective in several trials, producing response rates of 30-52 % in patients with pretreated metastatic breast cancer. To improve on tolerability and handling of the regime carboplatin may be the more appropriate choice for treatment. The mechanism of action of carboplatin is very similar to that of cisplatin. The rational for combining gemcitabine and carboplatin is based on their single-agent activities in metastatic breast cancer, the activity of this combination in other malignancies and on the fact that carboplatin has demonstrated efficacy comparable with cisplatin in several tumor types.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic breast cancer
* All patients were required to give written informed consent.
* Prior treatment with chemotherapy, hormonal therapy, immunotherapy or local radiotherapy was allowed (except gemcitabine or platinum agents).
* Patients were required to have at least one bidimensionally measurable lesion outside a previous radiation port.
* Age ≥ 18 years
* Karnofsky Performance status ≥ 70 %
* Minimal life expectancy of 12 weeks
* Adequate haematological, renal, cardiac and hepatic function:

  1. Leukocyte count ≥ 3.0 x 109/l
  2. Absolute neutrophil count ≥ 2.0 x 109/l
  3. Platelet count ≥ 100 x 109/l
  4. Haemoglobin ≥ 8 g/dl
  5. Total serum bilirubin ≤ 1.25 x upper limit of normal (ULN) In presence of liver metastasis ≤ 3 x ULN
  6. Transaminase (ALT,AST) level ≤ 3 x ULN In presence of liver metastasis ≤ 5 x ULN
  7. Alkaline phosphatase level ≤ 2.5 x ULN
  8. Creatinine clearance was required to exceed 60 ml/min.

Exclusion Criteria:

* Prior treatment with gemcitabine or platinum agents
* Inadequate creatinine clearance (< 60 ml/min)
* Only bone metastases
* Symptomatic brain metastases
* Women who are pregnant, lactating or refuse effective contraception
* Secondary malignancy
* History of another primary malignant disease other than in situ carcinoma of the uterine cervix or adequately treated basal cell skin cancer
* Active infection
* Any other concomitant severe clinical condition making implementation of the protocol including pre-hydration difficult.

Ages: 18 Years to 75 Years | Sex: Female
Age Groups: Adult, Older Adult
Dates: Start 2004-03; Study Completion 2006-10

CONTACTS AND LOCATIONS:
Overall Officials: Volker Heinemann, MD, Principal Investigator — University of Munich - Klinikum Grosshadern